CLINICAL TRIAL: NCT05601843
Title: Use of Transcutaneous Electrical Nerve Stimulation (TENS) for Acute Low Back Pain in the Emergency Department
Brief Title: Transcutaneous Electrical Nerve Stimulation for Back Pain in the Emergency Department (TENS-ED)
Acronym: TENS-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sam Brophy (Other)
Responsible Party: Sponsor-Investigator, Sam Brophy, Principal Investigator, Vancouver Island Health Authority
Organization: Vancouver Island Health Authority (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H21-02812
Record Dates: First submitted 2022-10-17; First posted 2022-11-01 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Back Pain; Muscle Pain; Acute Pain; Lower Back Pain; Lower Back Pain Mechanical
Keywords: Back pain; Mechanical back pain; Lower back pain; TENS; Transcutaneous Electrical Nerve Stimulation; Emergency; Emergency Department; Acute pain
MeSH Terms: conditions — Back Pain; Myalgia; Acute Pain; Low Back Pain; Emergencies | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TENS Arm (Experimental): Participants randomized to receive treatment with TENS in addition to standard care.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Control Arm (No Intervention): Participants randomized to not receive treatment with TENS. These participants receive standard care only.

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — TENS pads will be applied in a frame pattern around the area of maximal pain, as pointed out by the patient. The pads will be no more than 6 cm and no less than 3 cm away from the subjective area of maximal pain. The frequency of the TENS machine will be set to 100 Hz and the patient will be instructed on how to increase and decrease the amplitude based on their comfort. The patient will also be instructed on how to turn off the machine if they wish for any reason. Research assistants will be standing by during the intervention period to intervene if the patient requires assistance with the device.
  Other Names: Impulse® 3000 T (© 2014 BioMedical Life Systems, Inc.)
  Arms: TENS Arm

SUMMARY:
The effectiveness of Transcutaneous Electrical Nerve Stimulation (TENS) to reduce pain scores for patients with acute back pain in an ambulatory emergency department (ED) population will be examined in this dual-center, cluster randomized, controlled, open-label study.

DETAILED DESCRIPTION:
Back pain is one of the top 5 most common ED presenting complaints, accounting for approximately 3% of all ED visits. It is estimated that 85% of these patients will leave the ED with a non-specific diagnosis, such as mechanical low back pain, and will recover within 4-6 weeks. Unfortunately, treatment for these patients is limited and often consists of NSAIDs, acetaminophen, and opioids if in significant pain.

TENS is a non-pharmacological option for the treatment of pain. The mechanism of its effect is based on the gate control theory of pain; stimulation of large, myelinated fibers reduces transmission of pain through smaller, nociceptive C-fibers through inhibitory actions of interneurons. It is very safe, with very few reported adverse effects and a short list of contraindications.

In 2015, a Cochrane review examined the benefit of TENS in acute pain, which was defined as less than 12 weeks. Their review demonstrated tentative evidence of benefit in reducing pain, although due to the small sample sizes of the encompassing trials and the inability to blind, definitive conclusions are impossible.

Research question: "In patients in the ED triage area,18 years of age or older with acute or acute-on-chronic back pain for less than three weeks, does 30 min of transcutaneous electrical nerve stimulation reduce pain scores as compared to standard care alone?"

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Acute or acute-on-chronic back pain, defined as less than 3 weeks of increased symptoms.
* Canadian Triage and Acuity Scale (CTAS) level 3-5 in ambulatory section of emergency department8.
* Projected wait-time of at least 30 minutes.
* Comfortable with communication in English. Unfortunately, currently, we do not have the capacity or funding to hire a translator to translate our study documents or communicate with potential study participants.

Exclusion Criteria:

* Back pain "red flags" on initial history. These include:

  * Patient reported fever.
  * Recent direct blunt or penetrating trauma to the back, perceived by the patient to be the cause of acute pain or exacerbation of chronic pain.
  * Bilateral radicular symptoms.
  * Changes in ability to empty bladder or urinary incontinence since onset of back pain.
  * Incontinence of stool.
  * Saddle anesthesia.
  * Intravenous drug use within the last 30 days.
* History of spinal cord injury.
* Epilepsy.
* Abnormal triage vital signs:

  * Temperature greater than 38 C
  * Abnormal blood pressure (BP) defined as systolic BP less than 90 or over 180.
  * Tachypnea with respiratory rate (RR) greater than 22.
* Active pregnancy (patient warning on product label)
* Canadian Triage and Acuity Scale (CTAS) level 1-2.
* Implanted pacemaker or neurostimulation device.
* TENS unit in use by another patient at time of screening
* Wound, abrasion, rash over where TENS pads will be placed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Pain Score Difference | Change from baseline score at 60 minutes of study participation.
  Pain score as a primary outcome will be assessed by determining the difference in VAS between T0 and T60. VAS is a validated tool for measuring subject reports of pain in a variety of patient care settings. T60 was chosen as the primary endpoint as this was thought to allow sufficient time for standard care (ie. pharmacotherapy) to take effect. A clinically significant reduction of pain was defined as 30% on VAS, based on prior literature.

SECONDARY OUTCOMES:
Pain score at T30 | After 30 minutes of study participation.
  As a secondary outcome, pain score reduction at T30 will be assessed. This is to determine how effective TENS is at reduction pain immediately when finishing treatment. Similarly, a 30% reduction of pain score is considered clinically significant. No further assessment points will be used due to the variability of wait-times and high likelihood of loss to follow-up with later assessment points. We currently do not have capacity for telephone follow-up the next day.
Opioid requirements | After 60 minutes of study participation.
  A further secondary outcome is opioid requirements while in the ED, calculated by Oral Morphine Equivalents (OMEs). The duration of 8 hours or at time of discharge was determined to be an adequate length of time to allow for appropriate up-titration of opioids to achieve adequate pain treatment. Other forms of analgesia (ie. NSAIDs and acetaminophen) will not be tallied, due to the challenge of reliably interpreting the data - most patients have taken some form of over-the-counter analgesia prior to their ED encounter and different NSAIDs are often used without a reliable way of determining comparable such as OMEs for opioids.
ED Return Visits | Within 2 weeks of study participation.
  Return visits to the ED within 2 weeks will also be compared between groups, specifically analyzing the proportion of repeat presentations with a triage complaint of "back pain." This will be done by accessing the EMR of each patient in the trial through by the PI or CIs. Presentations to all EDs in the Island Health region are available upon accessing our local EMR (PowerChart). No further details other than initial triage complaint will be collected on these repeat visits.

OTHER OUTCOMES:
Adverse effects | Immediately after intervention.
  Adverse effects will also be gathered, including skin irritation and pad removal due to discomfort. Any other suspected adverse events will be recorded and reported in a narrative format.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Brophy, Principal Investigator — Island Health
Locations (1):
- Royal Jubilee Hospital, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No